CLINICAL TRIAL: NCT02130570
Title: Relative Patient Benefits of a Hospital-PCMH Collaboration Within an ACO to Improve Care Transitions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jeffrey L. Schnipper, MD.,MPH., Associate Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: 2012P000096
Record Dates: First submitted 2014-05-01; First posted 2014-05-05 (Estimated); Results first posted 2019-08-20 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Adverse Events; Readmissions; Patient Engagement
Keywords: Adverse events; Readmissions; Patient Centered Medical Home (PCMH); Accountable Care Organizations (ACO); Medication reconciliation; Discharge Advocate; Patient engagement; Transitions of care; Transitions coach; Pharmacist intervention
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Intervention Model Description: This is a stepped-wedge design, where each primary care practice starts in usual care, and then at a randomly selected point in time switches to the intervention arm.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multi-Model Intensive Discharge Program (Experimental): Multi-Model Intensive Discharge Program
  Interventions: Other: Multi-Model Intensive Discharge Intervention
- Usual Care (No Intervention): Usual Care

INTERVENTIONS:
Other: Multi-Model Intensive Discharge Intervention — 1. Inpatient medication safety interventions
  2. Inpatient "discharge advocate"
  3. Structured visiting nurse (VNA) appointments
  4. Post-discharge phone call by primary care personnel within 2 business days of discharge
  5. Structured post-discharge clinic appointment with PCP and other PCMH personnel within 2 weeks of discharge
  6. Improved communication between inpatient and primary care teams
  7. High-risk patients will receive additional interventions as needed:
     1. Home pharmacist visit
     2. Enrollment in the Partners integrated Care Management Program (iCMP)
     3. Enrollment in telemedicine programs for patients with CHF
     4. Palliative care consultation regarding goals of care
  8. Novel health information technology to facilitate communication and transfer of clinical information
  Arms: Multi-Model Intensive Discharge Program

SUMMARY:
The objective of this study is to design and implement a set of procedures (the intervention) to improve patients' experiences when they are discharged home from the hospital. Second, this study aims to look at how the intervention affects problems that are known to occur after discharge, including medication issues, worsening medical problems, or readmission to the hospital. The investigators will study how well patients recover the ability to do the things they could before they were admitted to the hospital and their opinions of the discharge process. Lastly, this study will look to understand the best way to implement the intervention into different hospitals and practices, and which types of patients benefit from it most.

DETAILED DESCRIPTION:
The specific aims of this study are:

1. To develop, implement, and refine a multi-faceted, multi-disciplinary transitions intervention with contributions from hospital and Patient-Centered Medical Home (PCMH) personnel.

   Hypothesis: a collaborative transitions intervention can be designed and implemented within an ACO that reliably provides the components of an ideal transition in care.
2. To evaluate the effects of this intervention on post-discharge adverse events, functional status, patient engagement, and emergency department and hospital utilization within 30 days of discharge.

   Hypothesis: compared with usual care, a collaborative transitions intervention will decrease post discharge adverse events, improve post-discharge functional status, increase patient engagement, and reduce emergency department and hospital utilization in the post-discharge period.
3. To understand barriers to and facilitators of successful implementation of this intervention across practices.

Hypothesis: several barriers to and facilitators of implementation can be identified and used to create lessons learned for other health systems to successfully implement this type of intervention.

ELIGIBILITY:
Inclusion Criteria:

Potential subjects will be adult patients admitted to medical and surgical services at BWH and MGH, likely to be discharged back to the community, and whose PCP belongs to one of the Partners Community Healthcare, Inc. (PCHI) primary care practices that has met "Primed" criteria for being a PCMH, admits at least 2 patients to BWH or MGH, and has agreed to participate. Primed criteria are a standard set of requirements that cover 6 essential building blocks of PCMH practices: electronic health record, patient portal, team-based care, practice redesign, care management, and identification of high-risk patients. We estimate that of the approximately 300 PCHI adult primary care practices, 150 of them will meet PCMH criteria during the study and that 20 of them will qualify and be willing to participate in the study. We estimate that 12,000 such patients will be admitted to BWH and MGH over the 18-month study period, of which we will enroll 1700 patients. These patients are broadly representative of hospitalized patients and include several vulnerable populations, including the elderly (33% 65 or older), patients with multiple chronic conditions (47% with Elixhauser comorbidity score 5 or more), and racial and ethnic minorities (14% African American, 13% Latino).

Exclusion Criteria:

1. Likely discharge to a location other than home (or to a caregiver's home)
2. Police custody
3. No telephone or homeless
4. Previous enrolment in the study
5. Patient unable to communicate in either English or Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1679 (Actual)
Dates: Start 2013-06; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L Schnipper, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
Voluntarily participating in PCORI's Open Science Pilot

RESULTS

PARTICIPANT FLOW:
Recruitment Details: BWH participants were enrolled from 8/21/2013 to 5/15/2015. MGH participants were enrolled from 9/18/2013 to 10/13/2015. Participants were recruited while they were inpatients on the medical or surgical services at either BWH or MGH.
Pre-assignment Details: A total of 141 eligible participants were enrolled to 1 pilot practice at Brigham and Women's Hospital and 1 pilot practice at Massachusetts General Hospital. These participants received the study Intervention so that we could troubleshoot and refine the Intervention procedures. These participants are NOT counted in the final enrollment number.
Groups:
- Usual Care: Patients receive the care that they would normally receive.
Period: Overall Study
Arm/Group | Multi-Model Intensive Discharge Program | Usual Care
Started | 987 | 692
Completed | 978 (Participants enrolled, did not die during index admission, did not withdraw consent) | 679 (Participants enrolled, did not die during index admission, did not withdraw consent)
Not Completed | 9 | 13
Not completed — Death | 3 | 5
Not completed — Withdrawal by Subject | 6 | 3
Not completed — Part of practice that discontinued study | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Usual Care: Patients receive the same care they would normally receive.
- Total: Total of all reporting groups
Arm/Group | Multi-Model Intensive Discharge Program | Usual Care | Total
Number analyzed (Participants) | 978 | 679 | 1657
Age, Customized [Number; unit: participants]
  Between 18 and 69 years | 700 | 477 | 1177
  >=70 years | 278 | 202 | 480
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 540 | 364 | 904
  Male | 438 | 315 | 753

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With an Adverse Event Within 30 Days After Index Discharge Date
Description: Proportion of Participants With an Adverse Event Within 30 Days after Index Discharge Date
Time Frame: 30 days after discharge
Population: 1679 participants were enrolled in the study, however, 22 patients were lost to follow-up and therefore not included in the analysis (e.g., patient withdrew consent, patient died during index admission).
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- Multi-Model Intensive Discharge Program: Multi-Model Intensive Discharge Program
  Multi-Model Intensive Discharge Intervention: 1. Inpatient medication safety interventions 2. Inpatient "discharge advocate" 3. Structured visiting nurse (VNA) appointments 4. Post-discharge phone call by primary care personnel within 2 business days of discharge 5. Structured post-discharge clinic appointment with PCP and other PCMH personnel within 2 weeks of discharge 6. Improved communication between inpatient and primary care teams 7. High-risk patients will receive additional interventions as needed:
  1. Home pharmacist visit
  2. Enrollment in the Partners integrated Care Management Program (iCMP)
  3. Enrollment in telemedicine programs for patients with CHF
  4. Palliative care consultation regarding goals of care 8. Novel health information technology to facilitate communication and transfer of clinical information
- Usual Care: Patients receive the care they would normally receive.
Arm/Group | Multi-Model Intensive Discharge Program | Usual Care
Number analyzed (Participants) | 978 | 679
proportion of participants | 0.18 [0.15 to 0.21] | 0.23 [0.20 to 0.27]
Statistical Analysis 1: Comparison: Multi-Model Intensive Discharge Program vs Usual Care; Test type: Superiority; p = 0.02, Regression poissant — This is the P-value for the adjusted IRR; Please see the "Other Statistical Analysis" field for adjustments; Incidence rate ratio = 0.52, 95% CI 2-sided [0.30 to 0.91]; Adjusted for study month, Elixhauser comorbidity score, patient age, sex, language, race/ethnicity, cognitive status, health literacy, functional status one month prior to admission, caregiver status, median income by zip code, ED visits in the previous 6 months, HOSPITAL readmission risk score, inpatient unit, and primary care practice. IRR: incidence rate ratio

2. Secondary Outcome: Proportion of Participants With New or Worsening Signs/Symptoms Within 30 Days of Discharge
Description: New or worsening signs or symptoms, i.e. unpleasant symptoms, loss of function, abnormal lab results, and/or additional medical care within 30 days after discharge.
Time Frame: 30 days after discharge
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Multi-Model Intensive Discharge Program | Usual Care
Number analyzed (Participants) | 978 | 679
proportion of participants | 0.90 [0.86 to 1.01] | 0.92 [0.85 to 0.97]
Statistical Analysis 1: Comparison: Multi-Model Intensive Discharge Program vs Usual Care; Test type: Superiority; p = 0.01, Regression poissant — This is the p-value for the adjusted rate; For adjustments, please see the "Other Statistical Analysis" field below; Incidence rate ratio = 0.78, 95% CI 2-sided [0.64 to 0.95]; [other analysis details as in outcome 1, analysis 1]

3. Secondary Outcome: Number of Patients With a Nonelective Readmission Within 30 Days of the Index Discharge Date
Description: Nonelective readmission within 30 days of the index discharge date
Time Frame: 30 days after discharge
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Multi-Model Intensive Discharge Program | Usual Care
Number analyzed (Participants) | 978 | 679
participants | 107 | 78
Statistical Analysis 1: Comparison: Multi-Model Intensive Discharge Program vs Usual Care; Test type: Superiority; p = 0.77, Regression, Logistic — This is the P-value for the adjusted Odds Ratio; For adjustments, please see the "Other Statistical Analysis" field below; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.64 to 1.85]; Adjusted for study month, Elixhauser comorbidity score, patient age, sex, language, race/ethnicity, cognitive status, health literacy, functional status one month prior to admission, caregiver status, median income by zip code, ED visits in the previous 6 months, HOSPITAL readmission risk score; clustered by inpatient unit; primary care practice as a random effect . OR: odds ratio

4. Secondary Outcome: Change in Functional Status on the Modified Medical Outcomes Survey Short Form-12 (SF-12v2) From One Month Prior to Admission to 30 Days After Discharge.
Description: During the inpatient enrollment period, patients will complete a modified Medical Outcomes Survey Short Form-12 (SF-12v2). The SF-12v2 measures a patient's functional status and health-related quality of life one month prior to admission. 30 days after discharge, SF12 questions will be repeated so that functional status and health-related quality of life can be compared to prior to admission.
  This measure is a 12-item measure. Each item 5 possible responses with a value from 1 to 5 (with higher scores indicating worse outcomes). A summary score is computed by summing the score on each item. Therefore, the range of summary scores for the SF-12v2 is a minimum of 12 and a maximum of 60.
Time Frame: One month prior to admission to 30 days after discharge.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Multi-Model Intensive Discharge Program | Usual Care
Number analyzed (Participants) | 978 | 679
units on a scale | 47.25 (7.85) | 46.14 (8.11)
Statistical Analysis 1: Comparison: Multi-Model Intensive Discharge Program vs Usual Care; Test type: Superiority; p = 0.91, Regression, Linear — This is the P-value for the adjusted difference; Please see the "Other Statistical Analysis" field for adjustments; Mean Difference (Final Values) = 0.08; Adjusted for study month, Elixhauser comorbidity score, patient age, sex, language, race/ethnicity, cognitive status, health literacy, functional status one month prior to admission, caregiver status, median income by zip code, ED visits in the previous 6 months, HOSPITAL readmission risk score; clustered by inpatient unit; primary care practice as a random effect

5. Secondary Outcome: Proportion of Participants With Positive Responses Regarding Patient Engagement and Opinions of the Discharge Process
Description: During the 30 day post-discharge follow-up phone call we asked patients about their participation in, understanding of, and ability to carry out the post-discharge plan. These questions include questions from the Interpersonal Processes of Care survey and several additional questions from the HOMERUN study of readmitted patients.
  In the table below, we have abbreviated each survey question since the number of characters is limited in this field in the table. We have pasted below the full survey question.
  1. When you were getting ready to leave the hospital one month ago, how often did your care team use medical terminology that you did not understand?
  2. How often did you feel confused about what was going on with your medical care because they did not explain things well?
  3. How often did they give you enough time to say what you thought was important regarding your medical care?
  4. How often did they listen carefully to what you had to say?
  5. How often did you feel p
Time Frame: 30 days after discharge
Population: 1679 participants were enrolled in the study, however, 22 patients were lost to follow-up and therefore not included in the analysis (e.g., patient withdrew consent, patient died during index admission). Not all patients answered the 30-day patient survey.
Measure: Number; unit: proportion of participants
Arm/Group | Multi-Model Intensive Discharge Program | Usual Care
Number analyzed (Participants) | 458 | 414
proportion of participants
  Used medical terminology you did not understand | .86 | .85
  Felt confused because things not explained well | .86 | .88
  Not given enough time to say what was important | .92 | .90
  How often did care team listen carefully to you | .94 | .92
  Felt pressured to have treatment not sure about | .95 | .95
  Asked if you might have problems w/ recommended tx | .41 | .34
  Understood what to do to care for self | .98 | .97
  Able to take medications correctly every day | .95 | .95
  Knew danger signs to watch and what to do | .96 | .94
  Knew how to contact my doctor if needed | .98 | .96
  Able to get to my doctor's appointment or tests | .95 | .95
  Able to follow diet team ordered for me | .41 | .52
  Had enough support from friends, family or others | .97 | .96
Statistical Analysis 1: Comparison: Multi-Model Intensive Discharge Program vs Usual Care; Test type: Superiority; p = 0.57, Regression, Logistic — Please see the "Other Statistical Analysis" field for adjustments and the P-value computed for each survey question; Odds Ratio, log = 0.85, 95% CI 2-sided [0.47 to 1.51] — Please see the "Other Statistical Analysis" field for a list of the estimated value and 95% CI for each survey question; Please see the "Other Statistical Analysis" field for adjustments

6. Secondary Outcome: Post-Discharge Health Care Utilization
Description: We will measure emergency department visits and hospital readmissions within 30 days of discharge using a combination of administrative data for all Partners hospitals plus patient report for all utilization outside the Partners system.
Time Frame: 30 days after discharge
Population: Post Discharge ED visits within 30 days of discharge were not able to be obtained from the second site MGH. Post discharge readmissions were obtained, however, without the ED visit data from MGH we are unable to create a count for Post-Discharge Health Care Utilization (ED plus readmissions).
Arm/Group | Multi-Model Intensive Discharge Program | Usual Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Multi-Model Intensive Discharge Program | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/978 | 0/679
Other Adverse Events (participants affected / at risk) | 0/978 | 0/679

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No